CLINICAL TRIAL: NCT06410274
Title: Ischaemic Lesions in Acute Intracerebral Haemorrhage: Pathophysiological Investigation Using Novel Multimodal Cerebral and Systemic Haemodynamic Assessments
Brief Title: Ischaemic Lesions in Acute Intracerebral Haemorrhage
Acronym: CHALLENGE-ICH
Status: Recruiting | Type: Observational
Sponsor: University of Leicester (Other)
Collaborators: University Hospitals, Leicester (Other)
Responsible Party: Sponsor
Other Study IDs: 0966
Record Dates: First submitted 2024-05-07; First posted 2024-05-13 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-04

CONDITIONS: Intracerebral Haemorrhage
Keywords: Stroke; Cerebral Autoregulation; Cerebral Blood Flow; Transcranial Doppler; Magnetic Resonance Imaging
MeSH Terms: conditions — Cerebral Hemorrhage; Stroke | interventions — Ultrasonography, Doppler, Transcranial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Intracerebral Haemorrhage Patients: Patients with a clinical diagnosis of haemorrhagic stroke on CT imaging within 48 hours of onset (for patients waking with a stroke, time of onset will be taken to be the time when the patient was last asymptomatic). This is a non-intervention study so no intervention will be given. However, the investigators will observe changes in cerebral haemodynamics of this group within 48 hours of stroke onset and within 3-7 days post-onset.
  Interventions: Device: Transcranial Doppler ultrasonography (TCD)

INTERVENTIONS:
Device: Transcranial Doppler ultrasonography (TCD) — TCD will be used to measure cerebral blood velocity (CBv) in the middle and posterior cerebral arteries (MCA and PCA). Following confirmation of a suitable TCD window, participants will undergo a ten-minute rest period in the supine or semi-supine position. Continuous measurements of CBv, blood pressure (BP), heart rate, and end-tidal carbon dioxide will be recorded. Baseline BP will be measured using an automated BP device prior to each recording to allow calibration of the files offline for analysis. This will occur at the first visit and at follow-up, 4-7 days post-onset of intracerebral haemorrhage.

SUMMARY:
The aim of this observational study is to determine how and why inadequate brain blood flow occurs after bleeding in patients with intracerebral haemorrhage (ICH). Treatment for strokes caused by burst blood vessels involves reducing blood pressure (BP) to stop the bleeding. However, this reduction in BP may affect blood flow, causing blockages in blood vessels within the brain. Fast breathing also affects brain blood flow. Therefore, participants will be asked to undergo a simple brain blood flow assessment using transcranial Doppler (TCD) within 48 hours upon admission to hospital. Patients will then have a follow-up TCD assessment at 4-7 days post-ICH onset, in addition to an MRI scan at >7 days. This research will help to confirm if blockages after bleeding are caused by reduced blood flow within the brain.

DETAILED DESCRIPTION:
Stroke is the second-leading cause of death worldwide, with high mortality and morbidity rates. One stroke type, intracerebral haemorrhage (ICH), refers to spontaneous, non-traumatic bleeding, within the brain tissue and is the second most common cause of stroke. Although ICH can happen at any age, it is more common over the age of 70. The most common cause of ICH is hypertension, which can cause bursting of cerebral blood vessels, resulting in bleeding within the brain. National and international guidelines strongly advocate systolic blood pressure (BP) lowering in ICH as part of "bundled" care, reducing fluctuations in cerebral blood velocity (CBv). However, despite blood pressure (BP) lowering being deemed clinically safe, no reduction in death or disability at 90 days was demonstrated in two landmark large randomised controlled trials. Moreover, reductions in BP may affect CBv to the whole of the brain, inadvertently causing ischaemic stroke (blockage of the blood supply).

Previous literature has identified that mild-to-moderate ICH stroke severity benefits from early and stable BP lowering, but those with excessively systolic high BP (>220 mmHg) prior to lowering suffer significantly higher rates of neurological deterioration. In order to understand the relationship between BP changes and potential clinical benefit in ICH, it needs to be determined if there is a global reduction in brain perfusion which is causing ischaemic lesions in the brain following ICH.

Prospective studies have shown impairments in dynamic cerebral autoregulation (dCA), cerebrovascular tone, and cerebrovascular resistance in acute ICH. Moreover, meta-analyses have demonstrated a previously unreported confounder to cerebral autoregulatory function: the presence of an acute reduction in spontaneous CO2 tension after ICH, potentially reflecting spontaneous hyperventilation (measured as partial pressure in arterial blood (pCO2) in patients in intensive care and on the ward). There is no current explanation for the presence of spontaneous hyperventilation post-ICH. However, it has been shown that across a range of end-tidal carbon dioxide (EtCO2) values, cerebral blood flow (CBF), dCA, and other core haemodynamic parameters (arterial BP and heart rate) have a dose-response relationship.

Fast breathing is also known to affect CBv. When EtCO2 is low, rapid acute cerebral vasoconstriction can occur - risking acute ischaemic injury. Therefore, in the presence of spontaneous hyperventilation or induced hyperventilation, reductions in brain perfusion through vasoconstriction could risk new or worsened ischaemic insults, particularly in the presence of BP lowering. Whilst the presence of cerebral small vessel disease plays a role in incidence of diffusion-weighted imaging (DWI) lesions after ICH, there have been no mechanistic association studies to date linking key confounding factors: BP lowering, EtCO2 change, dCA, and ischaemic lesions.

The investigators aim to perform transcranial Doppler (TCD) to measure CBv in patients with ICH within 48 hours of admission to hospital. These patients would then have a follow-up TCD assessment at 4-7 days post-ICH onset, in addition to a magnetic resonance imaging (MRI) scan (>7 days). Data would be collected and analysed to determine the relationship between cerebral haemodynamics and ischaemic lesions on MRI, post-acute ICH.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of a haemorrhagic stroke on CT imaging within 48 hours of onset (for patients waking with a stroke, time of onset will be taken to be the time when the patient was last asymptomatic).
* Male or female, aged 18 years or above.

Exclusion Criteria:

* MRI imaging is contraindicated or unlikely to tolerate scanning process due to clinical instability (GCS <8, unable to lie supine).
* Patients requiring anaesthesia.
* Male or Female, aged under 18 years.
* Clinical diagnosis of stroke greater than 48 hours from onset

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The participants will be recruited from the Leicester Royal Infirmary stroke wards.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2029-01-31 (Estimated); Study Completion 2029-01-31 (Estimated)

PRIMARY OUTCOMES:
Cerebral blood velocity measurements within 48 hours of admission to hospital and 4-7 days after onset in intracerebral haemorrhage patients. | From enrolment to the end of the follow-up (7 days).
  Absolute values (cm/s) in cerebral blood velocity measurements in intracerebral haemorrhage patients.
Cerebral blood velocity measurements within 48 hours of admission to hospital and 4-7 days after onset in intracerebral haemorrhage patients. | From enrolment to the end of the follow-up (7 days).
  Percentage change (%) in cerebral blood velocity measurements in intracerebral haemorrhage patients.
End-tidal carbon dioxide measurements within 48 hours of admission to hospital and 4-7 days after onset in intracerebral haemorrhage patients. | From enrolment to the end of the follow-up (7 days).
  Absolute values (mmHg) in end-tidal carbon dioxide measurements in intracerebral haemorrhage patients.
End-tidal carbon dioxide measurements within 48 hours of admission to hospital and 4-7 days after onset in intracerebral haemorrhage patients. | From enrolment to the end of the follow-up (7 days).
  Percentage change (%) in end-tidal carbon dioxide measurements in intracerebral haemorrhage patients.

SECONDARY OUTCOMES:
Arterial spin labelling magnetic resonance imaging measurements >7 days post-intracerebral haemorrhage onset. | From enrolment to the magnetic resonance imaging scan (<7 days post-intracerebral haemorrhage onset).
  Absolute values (mL/g/min) in arterial spin labelling magnetic resonance imaging measurements of cerebral blood velocity in response to a respiratory challenge.
Arterial spin labelling magnetic resonance imaging measurements >7 days post-intracerebral haemorrhage onset. | From enrolment to the magnetic resonance imaging scan (<7 days post-intracerebral haemorrhage onset).
  Percentage change (%) in arterial spin labelling magnetic resonance imaging measurements of cerebral blood velocity in response to a respiratory challenge (mL/g/min).

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospitals of Leicester NHS Trust, Leicester, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Individual patient data will not be shared, however once analysed and combined (statistically through mean averages etc), the results will be compiled into a report and submitted to a relevant journal, allowing researchers to view them.